CLINICAL TRIAL: NCT06779084
Title: Association Between Different Fasting Durations Before Bronchoscopy And The Discomfort Levels Of Patients Around The Procedure
Brief Title: Fasting Durations Before Bronchoscopy And The Discomfort Levels Of Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202412025RINA
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Bronchoscopy; Fasting ( 6H for Solid ; 2H for Clear Fluid )
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contemporary fasting principle (Experimental)
  Interventions: Other: contemporary fasting principle
- conventional fasting time (Active Comparator)
  Interventions: Other: conventional fasting time

INTERVENTIONS:
Other: contemporary fasting principle — (clear fluids for up to 2 hours before anesthesia)
  Arms: contemporary fasting principle
Other: conventional fasting time — (≥ 8 hours)
  Arms: conventional fasting time

SUMMARY:
The goal of this clinical trial is to learn if patients feel more comfortable while being placed on contemporary fasting principle than on conventional fasting time during flexible bronchoscopy. The main questions it aims to answer are:

To compare the thirty levels between patients with conventional fasting time (≥ 8 hours) and those with contemporary fasting principle (clear fluids for up to 2 hours before anesthesia) during flexible bronchoscopy To compare the levels of mucosal dryness between two groups of patients during flexible bronchoscopy To compare the levels of hunger between two groups of patients during flexible bronchoscopy To compare the levels of tiredness between two groups of patients during flexible bronchoscopy To compare the levels of fatigue between two groups of patients during flexible bronchoscopy To compare the levels of nausea/vomiting between two groups of patients during flexible bronchoscopy

Participants will:

Being placed on fasting either using conventional fasting time (≥ 8 hours) or with contemporary fasting principle (clear fluids for up to 2 hours before anesthesia) Being asked to respond to questions regarding thirsty, mucosal dryness, hunger, tiredness, fatigue, and nausea/vomiting in a visual analogue scale of 0 to 10

ELIGIBILITY:
Inclusion Criteria:

* planned flexible bronchoscopy

Exclusion Criteria:

* tracheostomy or intubated
* known to be pregnant
* significant functional or structural abnormalities of the gastrointestinal tract
* oral intake prohibited and infeasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
patient thirty level | right before the bronchoscopy procedure
  using a visual analogue scale of 0 to 10

SECONDARY OUTCOMES:
patient mucosal dryness | right before the bronchoscopy procedure
  using a visual analogue scale of 0 to 10
patient hunger | right before the bronchoscopy procedure
  using a visual analogue scale of 0 to 10
patient tiredness | right before the bronchoscopy procedure
  using a visual analogue scale of 0 to 10
patient fatigue | right before the bronchoscopy procedure
  using a visual analogue scale of 0 to 10
patient nausea | right after the bronchoscopy procedure
  using a visual analogue scale of 0 to 10
patient vomiting | right after the bronchoscopy procedure
  absent or present

IPD SHARING:
Plan to Share IPD: Undecided